CLINICAL TRIAL: NCT05426109
Title: Exploring the Role of Peanuts in Enhancing Healthy Weight Gain in Athletic Individuals
Brief Title: Role of Peanuts in Healthy Weight Gain in Athletic Individuals
Acronym: mGAINS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Responsible Party: Principal Investigator, Dawnine Enette Larson-Meyer, Professor, Virginia Polytechnic Institute and State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-561
Record Dates: First submitted 2022-06-15; First posted 2022-06-21 (Actual); Results first posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-05

CONDITIONS: Weight Gain
Keywords: Hypercaloric diet; Weight training; Lean mass; Body composition
MeSH Terms: conditions — Weight Gain

STUDY DESIGN:
Masking Description: Both the investigators and participants are aware of the group assignment since the foods prepared and provided (peanut-containing or no peanut snacks) cannot be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peanut snacks (Experimental): Participants will be provided and consume an extra 500 kcal/day of peanut-containing snacks for 10 weeks.
  Interventions: Other: Peanut snacks
- No peanut-containing snacks (Active Comparator): Participants will be provided and consume an extra 500 kcal/day of snacks without peanuts or peanut-containing foods for 10 weeks.
  Interventions: Other: No peanut-containing snacks

INTERVENTIONS:
Other: Peanut snacks — Participants will undergo a 10-week diet and weight training regimen to promote healthy weight gain. These participants will receive seven 500 kcal peanut-containing (whole peanuts or peanut butter) snacks each week and consume one snack per day throughout the study. They will also perform a series of weight training exercises supervised by a personal trainer on 3 days per week.
  Arms: Peanut snacks
Other: No peanut-containing snacks — Participants will undergo a 10-week diet and weight training regimen to promote healthy weight gain. These participants will receive seven 500 kcal non-peanut-containing high carbohydrate snacks each week and consume one snack per day throughout the study. They will also perform a series of weight training exercises supervised by a personal trainer on 3 days per week.
  Arms: No peanut-containing snacks

SUMMARY:
Many athletes and military personnel desire weight gain primarily as lean mass to improve performance and effectiveness in military/sport endeavors. While much is known about the energy restriction required to reduce body weight, very little is understood about energy and macronutrients needed to promote healthy gains in body weight and lean mass. Typically, athletes are encouraged to increase calorie intake by ~500 kcal/day with an emphasis on adequate protein and carbohydrate, and judicious inclusion of healthy fat-containing calorically-dense foods, including peanuts and peanut butter. This study proposes to evaluate the effect of a 10-week diet and exercise regimen designed to promote healthy weight gain. This will include increasing energy intake by 500 additional kcal/day (above weight maintenance diet) through daily provision of either peanut-based whole foods/snacks (peanut group) or a similar, high-carbohydrate, peanut-free snack (control group) along with a supervised strength training regimen. Results will serve as an important first step in helping understand the gaps in knowledge related to healthy weight gain, designing better weight gain meal plans, not only in athletes and military personnel, but also in clinical populations where promotion of weight gain is advocated.

ELIGIBILITY:
Inclusion Criteria:

* Interested in gaining 5 pounds of body weight to enhance effectiveness in sport, fitness, or military training/competition.
* Willing to eat 500 kcal/d and weight train 3x/wk for 10 weeks
* Have weight trained in the past 12 months
* Not taking medications or dietary supplements that influence study results
* Non-smoker
* Without any major medical problems (including high blood pressure or coronary heart disease)

Exclusion Criteria:

* Nut, peanut, tree nut or legume allergy
* No weight training experience
* Orthopedic limitations that affect ability to weight train
* Currently taking dietary supplements or prescribed pharmacological agents that may affect lean tissue accretion
* Current or past anabolic steroid use
* Have a history of or current signs of disordered eating
* Pregnant
* Abnormal levels of thyroid stimulating hormone or hemoglobin, serum lipids (e.g., fasting triglycerides >150 mg/dL and/or total cholesterol >200 mg/dL)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2021-11-22 (Actual); Primary Completion 2022-11-10 (Actual); Study Completion 2024-11-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Enette Larson-Meyer, PhD, Principal Investigator — Virginia Polytechnic Institute and State University
Locations (1):
- Virginia Polytechnic Institute and State University, Blacksburg, Virginia, United States

REFERENCES:
- [Derived] Sanchez AD, Reynolds JC, Marinik EL, Kolb RD, Lozano AJ, Davy BM, Hunter GR, Larson-Meyer DE. A Randomized Trial of Healthy Weight Gain in Athletic Individuals. Med Sci Sports Exerc. 2024 Aug 1;56(8):1454-1466. doi: 10.1249/MSS.0000000000003427. Epub 2024 Mar 23. PMID 38537251

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Peanut Snacks | No Peanut-containing Snacks
Started | 16 | 17
Completed | 16 | 16
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Peanut Snacks | No Peanut-containing Snacks | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Continuous [Median (Full Range); unit: years] — Population: Only included participants who completed the 10 wk intervention
  years | 23 [19 to 39] | 22 [18 to 28] | 23 [18 to 39]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Only including participants who completed the 10 week intervention
  Participants
    Female | 6 | 7 | 13
    Male | 10 | 9 | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Reported Race: Asian | 1 | 0 | 1
  Reported Race: White | 12 | 12 | 24
  Reported Race: Black/African American | 1 | 0 | 1
  Reported Race: Hispanic/Latino | 2 | 2 | 4
  Reported Race: Mixed (≥2 race categories) | 0 | 2 | 2
Total Body Mass [Mean (Standard Deviation); unit: kg] — Population: Only including participants who completed the 10-week intervention
  kg | 67.7 (12.7) | 70.4 (10.1) | 69 (11.4)

OUTCOME MEASURES:

1. Primary Outcome: Change in Total Body Mass (Weight)
Description: Participants will be weighed on a digital scale wearing standardized lab clothes at all scheduled testing sessions throughout the study.
Time Frame: 1-min laboratory measurement assessed at the baseline, 3-wk, 7-wk, and 11-week test sessions.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Peanut Snacks | No Peanut-containing Snacks
Number analyzed (Participants) | 16 | 16
kg
  11-wk | 1.6 (1.1) | 2.7 (1.2)
  7-wk | 1.8 (0.2) | 2.2 (0.1)
  3-wk | 0.8 (0.4) | 1.2 (0.3)

2. Primary Outcome: Change in Lean Body Mass
Description: Participants will undergo a dual-energy x-ray absorptiometry scan wearing standardized lab clothing at all scheduled testing sessions throughout the study. The scan analysis provides body composition results, including lean (fat-free) mass (kg).
Time Frame: 10-min laboratory measurement assessed at the baseline, 3-wk, 7-wk and 11-week test sessions.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Peanut Snacks | No Peanut-containing Snacks
Number analyzed (Participants) | 16 | 16
kg
  11-wk | 1.2 (1.1) | 1.9 (1.0)
  7-wk | 1.5 (0) | 1.7 (0)
  3-wk | 0.8 (0.4) | 1.1 (0.3)

3. Secondary Outcome: Change in Resting Metabolic Rate
Description: Participants will undergo a resting metabolic rate (RMR) test during select testing sessions throughout the study. The indirect calorimetry test measures the daily energy expenditure (or number of kilocalories needed to perform and maintain daily bodily functions) of each participant based on the measured gas exchange during the test.
Time Frame: 60-min laboratory measurement assessed at the baseline, 3-week, and 11-week test sessions.
Measure: Mean (Standard Error); unit: kcal/day
Arm/Group | Peanut Snacks | No Peanut-containing Snacks
Number analyzed (Participants) | 16 | 16
kcal/day
  11-wk | 1627 (369) | 1717 (338)
  3-wk | 1595 (253) | 1706 (258)
  BSL | 1541 (285) | 1632 (262)

4. Secondary Outcome: Change in Testosterone Levels
Description: Participants will have their blood collected by venipuncture in aseptic conditions. Testosterone (free) will be measured to determine the impact of the extra daily 500 kcal snacks on anabolism and muscle growth.
Time Frame: 5-min laboratory measurement assessed at the baseline, 3-week, 7-week, and 11-week test sessions.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Peanut Snacks | No Peanut-containing Snacks
Number analyzed (Participants) | 16 | 16
pg/mL
  11-wk | 18.5 (10.7) | 20.0 (10.3)
  7-wk | 19.0 (10.2) | 20.9 (9.8)
  3-wk | 18.5 (9.5) | 21.4 (11.3)
  baseline | 21.7 (9.7) | 23.5 (11.9)

5. Secondary Outcome: Change in Insulin-Like Growth Factor Levels
Description: Participants will have their blood collected by venipuncture in aseptic conditions. Insulin-like growth factor (IGF) will be measured to determine the impact of the extra daily 500 kcal snacks on anabolism and muscle growth.
Time Frame: 5-min laboratory measurement assessed at the baseline, 3-week, 7-week, and 11-week test sessions.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Peanut Snacks | No Peanut-containing Snacks
Number analyzed (Participants) | 16 | 16
ng/mL
  11-wk | 51.3 (21.4) | 53.4 (13.7)
  7-wk | 51.1 (17.4) | 49.4 (21.5)
  3-wk | 47.9 (20.2) | 45.0 (16.4)
  baseline | 49.8 (16.4) | 49.6 (14.2)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Peanut Snacks | No Peanut-containing Snacks
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-11-12): https://cdn.clinicaltrials.gov/large-docs/09/NCT05426109/Prot_SAP_000.pdf